CLINICAL TRIAL: NCT02958787
Title: Vessel Sparing Prostate Radiation Therapy: Dose Limitation to Critical Erectile Structures (Corpus Cavernosum and Internal Pudendal Artery) by MRI Based Treatment Planning
Brief Title: Vessel Sparing Prostate Radiation Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2004-0626
Record Dates: First submitted 2016-10-28; First posted 2016-11-08 (Estimated); Results first posted 2018-03-05 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-02

CONDITIONS: Cancer of the PROSTATE
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Vessel Sparing Radiation Therapy using MRI based treatment planning to limit dose to critical erectile structures
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — Radiation Therapy Using MRI Based Treatment Planning

SUMMARY:
Prostate cancer patients have a number of excellent treatment options to consider, and quality of life following treatment is often a consideration in treatment choice. One critical quality of life concern for patients diagnosed with prostate cancer is sexual function. Previous studies point to a vascular mechanism of impotence post-radiation therapy, as opposed to a nerve-based mechanism following surgery. In this study, the critical vascular structures (internal pudendal artery and corpus cavernosum) are defined by MRI-based imaging and included in treatment planning for radiation treatments, hopefully preserving critical artery function. This study will collect erectile function preservation rates at 5-years post-vessel-sparing radiotherapy with or without aids using the patient reported using the simplified three-question erectile function scale.

DETAILED DESCRIPTION:
The vast majority of patients diagnosed with prostate cancer in the modern era of PSA screening have localized and potentially curable disease. Patients have a number of excellent treatment options to consider, and quality of life following treatment is often a consideration in treatment choice. One critical quality of life concern for patients diagnosed with prostate cancer is sexual function. Studies of sexual function post-radiation therapy fall into three categories: incidence studies; correlative (dose and toxicity) studies; mechanism(functional) studies. All these studies point to a vascular mechanism of impotence post-radiation therapy, as opposed to a nerve-based mechanism following surgery. In this study, the critical vascular structures (internal pudendal artery and corpus cavernosum) are defined by MRI-based imaging and included in treatment planning for radiation treatments. Investigators propose that this technique will improve quality of life, sexual function, and relapse-free survival.

This study's primary aim is to determine erectile function preservation rates at 5-years post-vessel-sparing radiotherapy with or without aids using the patient reported using the simplified three-question erectile function scale.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of prostate cancer
* Patients must have measurable erectile function. Patients with erectile function on Viagra and drugs of the same class are eligible. Patients who require 6 months of hormonal therapy or less are eligible, provided baseline erectile function is measured prior to or within 14 days of the start of hormonal therapy.
* Baseline PSA (Prostate Specific Antigen), TNM stage (a classification of malignant tumors in cancer), and Gleason Score (A system of grading prostate cancer tissue based on how it looks under a microscope): Patients with low (PSA less than 10, T2a or less, Gleason 6 or less), intermediate, or high (Gleason 8-10, T3a, PSA over 20) risk disease are eligible for this protocol. Patients on finasteride or drugs of the same class are eligible.
* Patients must be 18 years or older. No upper age restriction.
* Patients treated with external beam radiotherapy alone or external beam therapy plus implant therapy are eligible.
* Patients must have an ECOG (Eastern Cooperative Oncology Group system of grading patient status that attempts to quantify cancer patients' general well-being and activities of daily life) performance status <2.
* The patient must sign study specific informed consent approved by the IRB of U of M indicating they are aware of the investigational nature of the treatment.

Exclusion Criteria:

* Patients who are impotent or have an IIEF (International Index of Erectile Function) <16.
* Patients who are medically ineligible for radiation therapy due to other medical conditions.
* Patients given hormonal therapy before baseline questionnaires filled out.
* Patients who receive implant only therapy.
* Patients unable to undergo MRI (Magnetic Resonance Imaging).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2004-11; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Spratt, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
No sharing

REFERENCES:
- [Derived] Spratt DE, Lee JY, Dess RT, Narayana V, Evans C, Liss A, Winfield R, Schipper MJ, Lawrence TS, McLaughlin PW. Vessel-sparing Radiotherapy for Localized Prostate Cancer to Preserve Erectile Function: A Single-arm Phase 2 Trial. Eur Urol. 2017 Oct;72(4):617-624. doi: 10.1016/j.eururo.2017.02.007. Epub 2017 Feb 21. PMID 28233591

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 135
Completed | 135
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 135
Age, Continuous [Median (Full Range); unit: years] | 63 [57 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 135

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients Able to be Sexually Active With or Without the Use of Aids
Description: The primary endpoint of the study was to accurately determine the preservation of erectile function post radiation therapy. Erectile preservation was defined as a score of 1 or 2 on the three-tier patient reported questionnaire equating to being able to be sexually active with or without aids.
  Scoring:
  1. Sexually active without aids
  2. Sexually active with aids
  3. Not sexually active with or without aids
Time Frame: 5 years from end of radiation treatment
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Intervention
Number analyzed (Participants) | 135
percentage of patients | 88 [81 to 92]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the length of the study, 5 years. The protocol was written to collect only adverse events relating to the intervention (questionnaire). The radiotherapy was given as standard of care and it was written that adverse events related to the standard of care treatment would not be collected.
Description: The protocol was written to collect only adverse events relating to the intervention (questionnaire). The radiotherapy was given as standard of care and it was written that adverse events related to the standard of care treatment would not be collected.
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/135
Serious Adverse Events (participants affected / at risk) | 0/135
Other Adverse Events (participants affected / at risk) | 0/135

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes